CLINICAL TRIAL: NCT04276116
Title: Effectiveness of the Evaluation and Communication of "Pulmonary Age" as Help for Smoking Cessation: a Cluster Randomized Essay
Brief Title: Effectiveness of the Evaluation and Communication of "Pulmonary Age" as Help for Smoking Cessation
Acronym: CAPAST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: APHP180456; 2019-A02060-57 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2020-01-31; First posted 2020-02-19 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Smoking Cessation
Keywords: smoking cessation; generally practice; pulmonary age; motivation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention)
- Usual care + communication of pulmonary age (Experimental)
  Interventions: Behavioral: Pulmonary age

INTERVENTIONS:
Behavioral: Pulmonary age — Communication of pulmonary age
  Arms: Usual care + communication of pulmonary age

SUMMARY:
The experimental design is a cluster randomized trial in 2 parallel groups: an intervention group with assessment of the pulmonary age and a control group without.

The population studied is patients aged 25 or more, smoking for more than a year, seen in general practice consultation, for any reason.

The progress of the study will be composed of an inclusion visit (M0) with a pulmonary age estimation for the intervention group and an measurement of the exhaled carbon monoxide for both groups, then a follow-up visit 6 months after the inclusion (M6) with an exhaled carbon monoxide measure for both groups, and a phone call at 12 months (M12) with a quality of life survey for both groups.

The primary outcome is the smoking cessation at 6 months, confirmed by the carbon monoxide exhaled, at a scheduled consultation with the General practitioner (GP).

DETAILED DESCRIPTION:
Few scientific studies evaluate the pharmacological and non-pharmacological measurement of pulmonary age for smoking cessation. Moreover, existing research studies provide contradictory results.

DESCRIPTION OF THE RESEARCH METHODOLOGY

Experimental design Cluster randomized controlled trial on the center (= medical practices) in 2 parallel groups (intervention group (pulmonary age estimation) and control group (no pulmonary age estimation)).

National multicentric research:

33 participating centers (= medical practices), located in France. 3 referring physicians (=regional coordinators) were identified to energize the team of investigators and facilitate inclusions. There are 3 in Ile de France and 1 in PACA.

Randomization

General practitioners who agree to participate in this study will be randomized according to a computerized procedure and centralized in 2 groups (=randomization in a cluster on the center (medical office)):

1. a group providing routine smoking cessation management (control group), which will not receive any specific guidance on the means to be used in this management.
2. a group providing routine smoking cessation management, accompanied by estimation and communication to the patient of the pulmonary age, measured using a PulmoLife electronic device. (Intervention Group)

Consenting patients will then receive smoking cessation assistance from their physician according to the randomization arm in which the physician is assigned (usual versus usual management + pulmonary age estimate and patient information). Patients will be called to the doctor's office 6 months later to measure the expired CO and complete a questionnaire on their tobacco consumption.

RESEARCH PROCESS

Patients will be invited to participate in the study by the general practitioner during a consultation, regardless of the reason for the consultation (tobacco-related or not)

Inclusion visit (M0)

During this visit, the inclusion and non-inclusion criteria will be verified. The general practitioner will present the study to the patient in detail (an information note on the study will have been given to him/her beforehand in the waiting room). If the patient agrees to participate in the study, his or her informed and written consent will be obtained.

The information collected by the general practitioner will be:

* socio-demographic data: age, sex, family situation, level of education, occupation, health insurance coverage (yes/no)
* overall health and co-morbidities
* smoking history: age of smoking onset, current number of cigarettes per day, average number of cigarettes since smoking began
* the number of withdrawal attempts, the maximum duration of withdrawal, the methods used, the date of the last attempt
* nicotine dependence (short Fagerström test), motivation to stop (Prochaska)
* chronic pathologies
* other addictions: collection of cannabis consumption
* respiratory symptoms (GOLD-CNAM questionnaire)
* overall health status (EQ-5D questionnaire)
* measurement of expired CO
* set of spirometric data from Pulmolife (FEV1, pulmonary age) (only for the "intervention" group) (= pulmonary age estimate)

It should be noted that whatever the group, the doctor will follow the patient according to current recommendations and his usual practice of managing smoking cessation.

6-month follow-up visit (+/- 15 days) (M6)

This visit will take place in both groups, 6 months +/- 15 days after the patient's inclusion.

During this visit, the doctor will collect:

* current smoking status (over the last 15 days)
* the measurement of expired CO
* the number of withdrawals attempts since inclusion, the duration of the attempts, the average number of cigarettes per day over the period
* the withdrawal assistance methods used during the period
* respiratory symptoms (GOLD-CNAM questionnaire)
* overall health status (EQ-5D questionnaire)
* intercurrent events
* the number of visits to the physician

  12 months visit (+/- 15 days) (M12)

During this visit (which will be made in the 2 groups of patients), will be collected by the doctor:

* Global health status data (EQ-ED)
* smoking status (over the last 15 days)
* the number of withdrawals attempts since inclusion, the duration of the attempts, the average number of cigarettes per day over the period
* the withdrawal assistance methods used during the period
* respiratory symptoms (GOLD CNAM questionnaire)
* intercurrent events
* the number of visits to the physician

This visit will correspond to the end of the patient's participation in the study.

EFFECTIVENESS EVALUATION

Description of efficacy evaluation parameters

The parameters for evaluating the effectiveness of the intervention are:

* Smoking cessation rate at 6 months from the intervention. Smoking cessation will be confirmed by measuring the exhaled CO at a scheduled 6-month follow-up consultation with the general practitioner
* Persistence of withdrawal at 12 months assessed by patient questionnaire: persistence of smoking cessation yes/no
* Smoking cessation rate at 12 months
* Characteristics of smoking cessation evaluated by questionnaire/patient:
* Smoking cessation yes/no, if no: reduction in tobacco consumption yes/no and number of cigarettes smoked per day at M6 versus M0
* Older smoking cessation for patients who have quit smoking
* Number of smoking cessation attempts within 6 months of the intervention and pharmacological and non-pharmacological measures implemented, including the use of alternative therapies (hypnosis, acupuncture, auriculotherapy, relaxation, etc.)
* Satisfaction of general practitioners measured by a satisfaction score on a Likert scale from 1 to 10

ELIGIBILITY:
Inclusion Criteria:

* Patient 25 years of age or older
* Smoker for a year or more
* Patient giving informed and written consent to participate in the study
* Patient affiliated to a social security scheme

Exclusion Criteria:

* Known respiratory illness, chronic or acute in progress or less than 3 weeks old (BPCO, asthma, other respiratory disease
* Refusal
* Myocardial infarction less than a year
* Chest or abdominal pain preventing or limiting completion of the forced exhalation maneuver necessary for evaluation of "pulmonary age", whatever the cause
* Oral or facial pain exacerbated by the mouthing of the mouthpiece
* Stress urinary incontinence
* Mental confusion or dementia
* Pregnant or breastfeeding woman
* Major protected
* Do not understand french

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2023-10-27 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Rate of smoking cessation at 6 months | 6 months
  assessed with carbon monoxide measure in exhaled air by ppm

SECONDARY OUTCOMES:
Assessment of tobacco cessation persistence at 12 months | 12 months
  Phone call
Tobacco cessation rate at 12 months | 12 months
  Phone call
Tobacco cessation characteristic | 6 months -12 months
  GP consultation-Phone call Survey
GP acceptability of the pulmonary age tool | 6 months
  assessed with the Likert scale (1-10)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Roche, MD, PhD, Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Saint Antoine, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Parkes G, Greenhalgh T, Griffin M, Dent R. Effect on smoking quit rate of telling patients their lung age: the Step2quit randomised controlled trial. BMJ. 2008 Mar 15;336(7644):598-600. doi: 10.1136/bmj.39503.582396.25. Epub 2008 Mar 6. PMID 18326503
- [Background] Lorenzo A, Noël F, Lorenzo M, Van Den Broucke J. Intérêt de la spirométrie en médecine générale pour la motivation au sevrage tabagique. Étude pilote de faisabilité et intérêt de l'" âge pulmonaire ".Rev Mal Respir. 13 févr 2017
- [Background] Kotz D, Wesseling G, Huibers MJ, van Schayck OC. Efficacy of confronting smokers with airflow limitation for smoking cessation. Eur Respir J. 2009 Apr;33(4):754-62. doi: 10.1183/09031936.00116308. Epub 2009 Jan 7. PMID 19129277
- [Background] Morris JF, Temple W. Spirometric "lung age" estimation for motivating smoking cessation. Prev Med. 1985 Sep;14(5):655-62. doi: 10.1016/0091-7435(85)90085-4. PMID 4070195